CLINICAL TRIAL: NCT06099886
Title: Repurposing Lithium as a Disease-modifying Therapy in Parkinson's Disease: A Phase I Trial
Brief Title: Repurposing Lithium for Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Thomas Guttuso, Principal Investigator, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007253; UL1TR001412 (NIH)
Record Dates: First submitted 2023-08-30; First posted 2023-10-25 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lithium aspartate (Experimental): Lithium aspartate capsules will be titrated in each patient to the maximum tolerated dosage between 30-45mg/day.
  Interventions: Dietary Supplement: Lithium aspartate

INTERVENTIONS:
Dietary Supplement: Lithium aspartate — Lithium aspartate 30-45mg/day
  Other Names: Lithitate

SUMMARY:
This study will examine the effects of lithium aspartate 30-45mg/day on MRI biomarkers and blood-based therapeutic targets among 15 early-stage Parkinson's disease patients.

DETAILED DESCRIPTION:
In observational studies, small daily doses of lithium have been associated with a 77% reduced risk of developing Parkinson's disease (PD). In addition, lithium therapy has been effective in preventing neuronal death and behavioral symptoms in several PD animal models. Recently, our group has shown 24-weeks of low-dose lithium aspartate therapy 45mg/day in PD to engage blood-based and the MRI disease progression biomarker, free water, to a greater extent than 15mg/day or 150mg/day of lithium carbonate. However, these blood-based and MRI biomarker findings stem from only four and two PD patients, respectively, who received lithium aspartate 45mg/day. In addition, two other PD patients receiving this dosage withdrew from the study due to side effects of sedation and dizziness. Subsequently, one of these patients who withdrew resumed lithium aspartate at 30mg/day and reported no side effects. Although these findings suggest that this dosage of lithium aspartate has positive effects on PD biomarkers, data from a larger number of PD patients will be required to justify conducting a larger, randomized controlled trial (RCT). The proposed study will enroll 15 additional PD patients over five months who will receive lithium aspartate 30-45mg/day for 24 weeks ensuring that the study will be completed within 12 months. The dosage will be slowly titrated in each patient up to the maximum tolerated dosage in this range. Blood-based biomarkers and MRIs will be assessed at baseline and 24 weeks. It is anticipated that a similar magnitude of biomarker engagement will be observed among these additional 15 patients as was seen in the handful from the pilot study. Such findings would provide strong preliminary evidence to support conducting a larger RCT including both clinical and biomarker outcomes. Positive results from such a RCT would support lithium aspartate as a disease-modifying therapy for PD.

ELIGIBILITY:
Inclusion Criteria:

Have PD for <4 years diagnosed by a movement disorder specialist. Have normal thyroid and renal function at the screening visit. Have no previous exposure to lithium therapy. Have no history of brain surgery. Have no hx of brain imaging findings suggesting another neurological condition besides PD.

Have no use of tobacco or THC products for >1 year. Have stable PD medications for >30 days without current need for adjustments in the investigator's opinion.

Have stable psychiatric and diuretic medications for >60 days with no anticipated need for changes for at least 24 weeks.

Have no active medical or psychiatric condition that may interfere with study procedures in the investigator's opinion.

Exclusion Criteria:

Have PD for >4 years or does not have PD. Have abnormal normal thyroid and renal function at the screening visit. Have previous exposure to lithium therapy. Have history of brain surgery. Have hx of brain imaging findings suggesting another neurological condition besides PD.

Have use of tobacco or THC products within the past year. Have PD medication adjustments within 30 days or needs PD medication adjustments in the investigator's opinion.

Have psychiatric or diuretic medication adjustments within the last 60 days or is anticipated to need changes over next 24 weeks.

Have active medical or psychiatric condition that may interfere with study procedures in the investigator's opinion.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
MRI-derived free water (FW) levels | Change from baseline (BL) to 24 weeks.
  FW in the posterior substantia nigra (pSN), dorsomedial nucleus of the thalamus (DMN-T) and the nucleus basalts of Meynert (nbM).
Peripheral blood mononuclear cell (PBMC) nuclear receptor-related 1 protein (Nurr1) mRNA expression. | Change from BL to 24 weeks.
  PBMC Nurr1 mRNA expression using Taqman PCR.

SECONDARY OUTCOMES:
Serum neurofilament light (NfL) | Change from BL to 24 weeks.
  Assessed using SIMOA platform
Serum glial fibrillary acidic protein (GFAP) | Change from BL to 24 weeks.
  Assessed using SIMOA platform
PBMC superoxide dismutase type-1 (SOD-1) mRNA expression | Change from BL to 24 weeks.
  PBMC SOD-1 mRNA expression using Taqman PCR.
PBMC pS9/total glycogen synthase kinase-3B (GSK-3B) ratio | Change from BL to 24 weeks.
  Assessed using ELISA
PBMC pThr308 and pS473/total protein kinase B (Akt) ratios | Change from BL to 24 weeks.
  Assessed using ELISA
Serum interleukin-6 | Change from BL to 24 weeks.
  Assessed using ELISA
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III (Motor Examination) | Change from BL to 24 weeks.
  Assessed in the "on" state. Score range 0-132 with higher scores indicating worse outcomes.
Montreal Cognitive Assessment (MoCA) | Change from BL to 24 weeks.
  Score range 0-30 with higher scores indicating better outcomes.
Parkinson's Anxiety Scale | Change from BL to 24 weeks.
  Score range 0-48 with higher scores indicating worse outcomes.
Geriatric Depression Scale-15 | Change from BL to 24 weeks.
  Score range 0-15 with higher scores indicating worse outcomes.
Fatigue Severity Scale | Change from BL to 24 weeks.
  Score range 9-63 with higher scores indicating worse outcomes.
Insomnia Severity Index | Change from BL to 24 weeks.
  Score range 0-28 with higher scores indicating worse outcomes.
Parkinson's Disease Questionnaire-8 | Change from BL to 24 weeks.
  Score range 0-32 with higher scores indicating worse outcomes.
Levodopa equilavent dose | Change from BL to 24 weeks.
  Higher scores indicate higher dose of dopaminergic therapy.

OTHER OUTCOMES:
Adverse events | Through study completion, an average of 24 weeks.
  Number of patients with serious adverse events and number who withdraw from the study.

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Williamsville, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will be considered on a case-by-case basis.

REFERENCES:
- [Background] Guttuso T Jr, Shepherd R, Frick L, Feltri ML, Frerichs V, Ramanathan M, Zivadinov R, Bergsland N. Lithium's effects on therapeutic targets and MRI biomarkers in Parkinson's disease: A pilot clinical trial. IBRO Neurosci Rep. 2023 May 7;14:429-434. doi: 10.1016/j.ibneur.2023.05.001. eCollection 2023 Jun. PMID 37215748